CLINICAL TRIAL: NCT01913223
Title: Endoscopic Sub-mucosal Dissection With the Nestis® Jet Injector System With a Bi-functional Catheter: First Prospective Trial.
Acronym: NESTIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011.709
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2014-08

CONDITIONS: Barrett's Esophagus; Intestinal Dysplasia; Esophageal Dysplasia; Colorectal Neoplasms
Keywords: Endoscopic submucosal dissection; jet injector; saline solution; safety; effectiveness
MeSH Terms: conditions — Barrett Esophagus; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- submucosal dissection by dissector water jet (Experimental)
  Interventions: Device: Nestis® jet injector system with a bi-functional catheter

INTERVENTIONS:
Device: Nestis® jet injector system with a bi-functional catheter

SUMMARY:
ESD (Endoscopic Sub-mucosal Dissection)is the first-intent method to treat superficial neoplasms of the digestive tract at it allows an en-bloc R0 resection. Following marking of the lesion margins, ESD comprises 3 steps: 1) liquid injection into the sub-mucosal space 2) circumferential (complete or partial) incision and 3) dissection of the submucosa. Several tools are necessary to perform ESD with the standard technique. Development of water jet with bi functional (injection and cutting) catheter allows time and significant reduction of perforation risk (due to multiple changes of instruments). For this purpose, Nestis introduced the Enki 2 pulsed jet technology with high pressure system to inject efficiently and at any time viscous solutions in direct viewing and retroflexion. Preliminary pig studies indicate that injection of glycerol, hyaluronate and hydroxyethlstarch with Enki 2 are possible. In addition, preclinical studies on living pig colon models using saline solutions have demonstrated that perforation rates and operating times are significantly reduced compared to a standard electrosurgical knife. The present clinical study is being performed to confirm this system capability to perform ESD in humans.

ELIGIBILITY:
Inclusion Criteria:

* in the esophagus: squamous cell carcinoma (well differentiated G1) or high grade dysplasia or neoplasia on barrett esophagus with high grade dysplasia or adenocarcinoma confirmed by two different pathologists, with only superficial tissue (mucosal invasion (T1m) and no lymph nodes on EUS endoscopy radial and mini probe), larger than 15 mm of diameter, with an extension of less than 10 cm high and less than two thirds of the esophageal circumference
* in the stomach: superficial adenocarcinoma or high grade dysplasia (well differentiated G1) with no depth invasion of the sub mucosa in EUS endoscopy and no lymph nodes according to the recommendations of the Japanese gastric cancer association, and with a diameter of more than 15 mm
* in the colon and the rectum: sessile serrated adenomas, adenomas or superficial adenocarcinoma (well differentiated G1), larger than 15 mm, corresponding to non granular Lateral spreading tumor (NG-LST) or granular (G-LST) with a focal Kudo V zone in the lesion, with a circumferential extension of less than two thirds and with only a superficial extension (no sub mucosal invasion and no lymph nodes in EUS endoscopy of the rectum).
* Consent form signed
* Anesthesiology risk limited with ASA score 1 or 2
* Patients over 18 years old
* Affiliation to social safety system

Exclusion Criteria:

* other lesions of the digestive tract
* high anesthetic risk (ASA score > 2)
* previous treatment of the lesion (radiotherapy, endoscopy, surgery, chemotherapy…)
* other malignant disease locally advanced or with metastasis
* hemostasis disorders
* pregnancy or breast feeding
* participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Safety outcome | At 1 month
  Safety is measured in term of perforation rate and bleeding rate with immediate complication or delayed one after the procedure, at one month complications are not linked to the ESD procedure

SECONDARY OUTCOMES:
Effectiveness of the procedure in terms of complete neoplasia resections | less than one month to get the pathology examination report
  Procedure is successful when the resection is complete with no residual tissue on the margins in depth and in the lateral part of the lesions.
Effectiveness of the procedure in terms of complete neoplasia resections | three month
  no macroscopic nor microscopic local recurrence during follow up endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Result] Pioche M, Lepilliez V, Ciocirlan M, Rivory J, Miaglia C, Hervieu V, Poncet G, Valette PJ, Saurin JC, Ponchon T. Endoscopic submucosal dissection with the Nestis(R) jet injector system with a bifunctional catheter: first prospective clinical trial (NCT: 2012-A00272-41). Surg Endosc. 2016 Nov;30(11):5140-5146. doi: 10.1007/s00464-016-4827-8. Epub 2016 Mar 4. PMID 26944726